CLINICAL TRIAL: NCT06488495
Title: A Randomized Controlled Trial on Exercise Program in Patients With Nontuberculous Mycobacterial Pulmonary Disease (NTM-Exercise)
Brief Title: Exercise Program in Patients With Nontuberculous Mycobacterial Pulmonary Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4-2024-0147
Record Dates: First submitted 2024-06-03; First posted 2024-07-05 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Nontuberculous Mycobacterial Pulmonary Disease
Keywords: NTM; Pulmonary Disease; Exercise
MeSH Terms: conditions — Lung Diseases; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Experimental): Participants receive the exercise intervention immediately after randomization
  Interventions: Behavioral: Exercise Program
- Delayed Intervention Group (Other): Participants receive the exercise intervention immediately after enrollment.
  Interventions: Behavioral: Exercise Program

INTERVENTIONS:
Behavioral: Exercise Program — The exercise intervention includes a six-week program with weekly supervised sessions and daily home-based exercises.
  Arms: Immediate Intervention Group
Behavioral: Exercise Program — The exercise intervention includes a six-week program with weekly supervised sessions and daily home-based exercises.
  Arms: Delayed Intervention Group

SUMMARY:
1.objective Evaluation of effectiveness and safety of exercise intervention program for patients with non-tuberculous mycobacterial pulmonary disease 2. background Nontuberculous mycobacterial pulmonary disease (NTM-PD) is a chronic respiratory infection that generally affects individuals with structural lung diseases, such as chronic obstructive pulmonary disease (COPD) and bronchiectasis and without structural lung disease. The prevalence of NTM-PD is increasing worldwide , which has caused public health concerns because of environmental exposure to nontuberculous mycobacteria (NTM) and chronic intractable diseases.

Pulmonary rehabilitation is essential to the non-pharmacological treatment of chronic respiratory diseases. Positive effects of exercise training have been demonstrated in COPD and bronchiectasis. However, there are limited data on the effectiveness and safety of exercise program for patients with non-tuberculous mycobacterial pulmonary disease 3. design

1) Prospective, single-center, randomized, open-label, two-group clinical study 2) Patients eligible for the study are randomly assigned 1:1 4. group

1. arm 1 : immediate exercise intervention group Exercise intervention will begin immediately after randomization.
2. arm 2 : delayed intervention group : Exercise intervention will begin 6 weeks after randomization.

5. intervention

1) 6-week exercise program : one-day hospital-based education, 5-day home-based exercise 6. Participants :

1) patients with nontuberculous mycobacterial pulmonary disease

* 40-80 years old
* culture positive within 6months
* with respiratory symptoms 7. Outcome measure

  1. primary outcome : Oxygen uptake max
  2. secondary outcome : 6MWT(six-minute walk test), quality of life, pulmonary function, body composition, inflammatory marker

DETAILED DESCRIPTION:
Background and Theoretical Basis

1. Necessity of Exercise Intervention in Patients with Nontuberculous Mycobacterial Pulmonary Disease NTM (Nontuberculous Mycobacteria) includes all mycobacterial species except for tuberculosis and leprosy bacteria. It is commonly found in water and soil, and the lungs are the most frequent infection site. NTM pulmonary disease is increasing globally and in Korea, where its incidence has risen almost fivefold from 11.4 per 100,000 in 2010 to 56.7 per 100,000 in 2021, surpassing the incidence of tuberculosis (52.1 per 100,000) in 2021.

   Economic Impact: Direct medical expenditures related to NTM pulmonary disease in Korea rapidly increased to 20.9 billion KRW in 2021, a 5.8-fold increase compared to 2010. Studies in Canada have shown that the average annual medical cost per NTM patient is $11,541, with higher costs associated with inpatient care prior to death. Reducing hospital admissions through improved prognosis via exercise interventions can be economically beneficial.

   Demographic Considerations: The incidence and mortality of NTM pulmonary disease are higher in those over 65 years old, with the prevalence rate being significantly higher in this age group (163.1 per 100,000 in 2021). With Korea's rapidly aging population, the prevalence and associated medical costs of NTM pulmonary disease are expected to increase.

   Clinical Considerations: NTM pulmonary disease has a long treatment period with frequent treatment failures and relapses. There is a need for adjunctive therapies beyond pharmacological treatment to improve patient prognosis. Studies have shown a correlation between muscle deterioration measured indirectly by CT and increased mortality in NTM patients, suggesting that exercise interventions to improve muscle quality could enhance patient outcomes.

   Conclusion: Developing an exercise intervention program as an adjunctive therapy may contribute to improving prognosis and quality of life for NTM pulmonary disease patients.
2. Recent Research Trends

Existing Research: There are few studies analyzing the effects of exercise interventions in NTM pulmonary disease patients. Two small-scale studies have been conducted on inpatient exercise interventions and chest physical therapy (using positive expiratory pressure devices or cough training). However, there is no large-scale study on outpatient exercise interventions.

Research Gaps: There is a lack of descriptive epidemiological studies on physical activity levels or muscle strength in NTM pulmonary disease patients, which are essential for setting appropriate exercise intervention goals. Existing studies on conditions frequently associated with NTM pulmonary disease, such as bronchiectasis or chronic obstructive pulmonary disease (COPD), have shown that exercise interventions can improve exercise capacity and quality of life.

Conclusion: Given the positive outcomes of exercise interventions in related conditions, further research on the effects of exercise interventions in NTM pulmonary disease patients is warranted.

4. Research Design

(1) Study Design

1. design

1) Prospective, single-center, randomized, open-label, two-group clinical study 2) Patients eligible for the study are randomly assigned 1:1

2. group

1. arm 1 : immediate exercise intervention group Exercise intervention will begin immediately after randomization.
2. arm 2 : delayed intervention group : Exercise intervention will begin 6 weeks after randomization.

3. intervention

1. 6-week exercise program : one-day hospital-based education, 5-day home-based exercise A structured exercise regimen tailored to each patient's physical capacity, including aerobic, resistance, and flexibility training, conducted over a 6-week period

4. Participants :

1. Incluison patients with nontuberculous mycobacterial pulmonary disease - 40-80 years old

   * culture positive within 6months
   * with respiratory symptoms
2. exclusion Patients with severe comorbid conditions, recent surgery, or those unable to participate in exercise programs

5. Procedure

* Baseline Assessment: All participants will undergo initial assessments, including medical history, physical examination, 6MWT, QOL, body composition, handgrip, and pulmonary function tests.
* Randomization: Participants will be randomly assigned to either the intervention group (immediate exercise group) or the control group (delayed exercise group) stratified by BACES score (low BACES (0/1) vs moderate to severe BACES (2-5))
* intervention : 6-week exercise program : one-day hospital-based education, 5-day home-based exercise A structured exercise regimen tailored to each patient's physical capacity, including aerobic, resistance, and flexibility training, conducted over a 6-week period
* Follow-up: Assessments will be repeated after 6-week program and 6 months later to evaluate the impact of the exercise intervention in the intervention group (immediate exercise program).

Assessments will be repeated after 6-week baseline examination, before exercise program and 6 months later to evaluate the impact of the exercise intervention in the control group (delayed exercise group)

Data Analysis: Statistical analyses will be performed to compare the outcomes between the intervention and control groups.

5. Ethical Considerations

Informed Consent: All participants will provide written informed consent before participation.

Ethical Approval: The study protocol was reviewed and approved by the institutional review board (IRB).

6. Outcome measure

1. primary outcome : VO2 max
2. secondary outcome : 6MWT, quality of life, pulmonary function, body composition, inflammatory marker

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40-80 diagnosed with NTM pulmonary disease.
* Present respiratory symptoms.
* Positive NTM culture within the last 6 months.
* Voluntary consent to participate.

Exclusion Criteria:

* Diagnosed with cardiovascular disease.
* Recent major hemoptysis.
* Musculoskeletal issues preventing free movement.
* Unable to read the consent form.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
VO2max, maximal oxygen consumption | Immediate intervention group : 1) before exercise program (baseline) 2) after 6-week exerrcise program 3) after 6 month of exercise program
  VO2max will be measured in baseline, after 6-week exercise program in the intervetion arm and baseline, before exercise program, and after 6-week exercise program in the control arm. The difference of VO2 max between the group will be assessed.

SECONDARY OUTCOMES:
physical function | Immediate intervention group : 1) Baseline (before exercise program), 2) Post-evaluation ( after 6-week exercise program), 3) long-term evaluation ( after 6months of exercise program)
  6min walk test will be measured in both intervention arm and control arm (delayed intervention group).
physical function | Delayed intervention group : 1) Baseline 2) Pre-evaluation (before exercise program), 3) Post-evaluation ( after 6-week exercise program), 4) long-term evaluation ( after 6months of exercise program)
  6min walk test will be measured in both intervention arm and control arm (delayed intervention group).
physical function | Immediate intervention group : 1) Baseline (before exercise program), 2) Post-evaluation ( after 6-week exercise program), 3) long-term evaluation ( after 6months of exercise program)
  30second sit to stand will be measured in both intervention arm and control arm (delayed intervention group).
physical function | Delayed intervention group : 1) Baseline 2) Pre-evaluation (before exercise program), 3) Post-evaluation ( after 6-week exercise program), 4) long-term evaluation ( after 6months of exercise program)
  30second sit to stand will be measured in both intervention arm and control arm (delayed intervention group).
physical function | Immediate intervention group : 1) Baseline (before exercise program), 2) Post-evaluation ( after 6-week exercise program), 3) long-term evaluation ( after 6months of exercise program)
  Short physical performance battery (SPPB) will be measured in both intervention arm and control arm (delayed intervention group).
physical function | Delayed intervention group : 1) Baseline 2) Pre-evaluation (before exercise program), 3) Post-evaluation ( after 6-week exercise program), 4) long-term evaluation ( after 6months of exercise program)
  Short physical performance battery (SPPB) will be measured in both intervention arm and control arm (delayed intervention group).
physical function | Immediate intervention group : 1) Baseline (before exercise program), 2) Post-evaluation ( after 6-week exercise program), 3) long-term evaluation ( after 6months of exercise program)
  global physical activity Questionnaire (GPAQ) : According to the GPAQ analysis guidelines, the metabolic equivalent of task (MET) min per week after assigning MET values (four METs for moderate intensity and eight METs for vigorous intensity) to incorporate the intensity of PA will be calculated. The score of less than 600 classifies the subject as inactive; a score of 600 or more classifies the subject as active.
physical function | Delayed intervention group : 1) Baseline 2) Pre-evaluation (before exercise program), 3) Post-evaluation ( after 6-week exercise program), 4) long-term evaluation ( after 6months of exercise program)
  global physical activity Questionnaire (GPAQ) : According to the GPAQ analysis guidelines, the metabolic equivalent of task (MET) min per week after assigning MET values (four METs for moderate intensity and eight METs for vigorous intensity) to incorporate the intensity of PA will be calculated. The score of less than 600 classifies the subject as inactive; a score of 600 or more classifies the subject as active.
Quality of Life | Immediate intervention group : 1) Baseline (before exercise program), 2) Post-evaluation ( after 6-week exercise program), 3) long-term evaluation ( after 6months of exercise program)
  Body composition will be measured by bioimpedance analysis using an InBody 770 device (Biospace, Seoul, Republic of Korea). Skeletal muscle mass, appendicular skeletal muscle mass, fat mass, fat free mass will be measured. Sarcopenia was diagnosed when patients also exhibited low appendicular skeletal muscle mass divided by height squared (<7.0 kg/m2 for males and <5.7 kg/m2 for females). Adipopenia was defined when the fat mass index (FMI) was below the lower limit of the normal range (<3 kg/m2 for males and <5 kg/m2 for females), based on a study examining normal FMI in a Korean population
Quality of Life | Delayed intervention group : 1) Baseline 2) Pre-evaluation (before exercise program), 3) Post-evaluation ( after 6-week exercise program), 4) long-term evaluation ( after 6months of exercise program)
  Body composition will be measured by bioimpedance analysis using an InBody 770 device (Biospace, Seoul, Republic of Korea). Skeletal muscle mass, appendicular skeletal muscle mass, fat mass, fat free mass will be measured. Sarcopenia was diagnosed when patients also exhibited low appendicular skeletal muscle mass divided by height squared (<7.0 kg/m2 for males and <5.7 kg/m2 for females). Adipopenia was defined when the fat mass index (FMI) was below the lower limit of the normal range (<3 kg/m2 for males and <5 kg/m2 for females), based on a study examining normal FMI in a Korean population
Quality of Life | Immediate intervention group : 1) Baseline (before exercise program), 2) Post-evaluation ( after 6-week exercise program), 3) long-term evaluation ( after 6months of exercise program)
  COPD assessment test (CAT) :The score will range from 0 to 40. Higher scores indicate COPD has a greater impact on the QOL.
Quality of Life | Delayed intervention group : 1) Baseline 2) Pre-evaluation (before exercise program), 3) Post-evaluation ( after 6-week exercise program), 4) long-term evaluation ( after 6months of exercise program)
  COPD assessment test (CAT) The score will range from 0 to 40. Higher scores indicate COPD has a greater impact on the QOL.
Quality of Life | Immediate intervention group : 1) Baseline (before exercise program), 2) Post-evaluation ( after 6-week exercise program), 3) long-term evaluation ( after 6months of exercise program)
  Quality of Life Questionnaire-Bronchiectasis (QOL-B) :Score will range from 0 to 100. Higher scores indicate COPD has a greater impact on the QOL. Higher scores indicate high QOL.
Quality of Life | Delayed intervention group : 1) Baseline 2) Pre-evaluation (before exercise program), 3) Post-evaluation ( after 6-week exercise program), 4) long-term evaluation ( after 6months of exercise program)
  Quality of Life Questionnaire-Bronchiectasis (QOL-B) : Score will range from 0 to 100. Higher scores indicate COPD has a greater impact on the QOL. Higher scores indicate high QOL.
Quality of Life | Immediate intervention group : 1) Baseline (before exercise program), 2) Post-evaluation ( after 6-week exercise program), 3) long-term evaluation ( after 6months of exercise program)
  Hospital anxiety and depression scale (HDAS) :The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). The scale distinguishes between mild symptoms (≥8) and severe symptoms (≥11) of depression or anxiety.
Quality of Life | Delayed intervention group : 1) Baseline 2) Pre-evaluation (before exercise program), 3) Post-evaluation ( after 6-week exercise program), 4) long-term evaluation ( after 6months of exercise program)
  Hospital anxiety and depression scale (HDAS) : The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). The scale distinguishes between mild symptoms (≥8) and severe symptoms (≥11) of depression or anxiety.
Pulmonary Function | Immediate intervention group : 1) Baseline (before exercise program), 2) Post-evaluation ( after 6-week exercise program), 3) long-term evaluation ( after 6months of exercise program)
  PFT(pulmonary function test)
Pulmonary Function | Delayed intervention group : 1) Baseline 2) Pre-evaluation (before exercise program), 3) Post-evaluation ( after 6-week exercise program), 4) long-term evaluation ( after 6months of exercise program)
  PFT(pulmonary function test)
Pulmonary Function | Immediate intervention group : 1) Baseline (before exercise program), 2) Post-evaluation ( after 6-week exercise program), 3) long-term evaluation ( after 6months of exercise program)
  FVC(forced vital capacity)
Pulmonary Function | Delayed intervention group : 1) Baseline 2) Pre-evaluation (before exercise program), 3) Post-evaluation ( after 6-week exercise program), 4) long-term evaluation ( after 6months of exercise program)
  FVC(forced vital capacity)
Pulmonary Function | Immediate intervention group : 1) Baseline (before exercise program), 2) Post-evaluation ( after 6-week exercise program), 3) long-term evaluation ( after 6months of exercise program)
  FEV1(forced expiratory
Pulmonary Function | Delayed intervention group : 1) Baseline 2) Pre-evaluation (before exercise program), 3) Post-evaluation ( after 6-week exercise program), 4) long-term evaluation ( after 6months of exercise program)
  FEV1(forced expiratory
Biochemical inflammatory marker | Immediate intervention group : 1) Baseline (before exercise program), 2) Post-evaluation ( after 6-week exercise program), 3) long-term evaluation ( after 6months of exercise program)
  CBC(complete blood count)
Biochemical inflammatory marker | Delayed intervention group : 1) Baseline 2) Pre-evaluation (before exercise program), 3) Post-evaluation ( after 6-week exercise program), 4) long-term evaluation ( after 6months of exercise program)
  CBC(complete blood count)
Biochemical inflammatory marker | Immediate intervention group : 1) Baseline (before exercise program), 2) Post-evaluation ( after 6-week exercise program), 3) long-term evaluation ( after 6months of exercise program)
  Albumin
Biochemical inflammatory marker | Delayed intervention group : 1) Baseline 2) Pre-evaluation (before exercise program), 3) Post-evaluation ( after 6-week exercise program), 4) long-term evaluation ( after 6months of exercise program)
  Albumin
Biochemical inflammatory marker | Immediate intervention group : 1) Baseline (before exercise program), 2) Post-evaluation ( after 6-week exercise program), 3) long-term evaluation ( after 6months of exercise program)
  CRP(C reactive protein)
Biochemical inflammatory marker | Delayed intervention group : 1) Baseline 2) Pre-evaluation (before exercise program), 3) Post-evaluation ( after 6-week exercise program), 4) long-term evaluation ( after 6months of exercise program)
  CRP(C reactive protein)
Biochemical inflammatory marker | Immediate intervention group : 1) Baseline (before exercise program), 2) Post-evaluation ( after 6-week exercise program), 3) long-term evaluation ( after 6months of exercise program)
  ESR(erythrocyte)
Biochemical inflammatory marker | Delayed intervention group : 1) Baseline 2) Pre-evaluation (before exercise program), 3) Post-evaluation ( after 6-week exercise program), 4) long-term evaluation ( after 6months of exercise program)
  ESR(erythrocyte)
Body composition and handgrip strength | Immediate intervention group : 1) Baseline (before exercise program), 2) Post-evaluation ( after 6-week exercise program), 3) long-term evaluation ( after 6months of exercise program)
  Body composition and handgrip strength be measured in both intervention arm and control arm(delayed intervention group).
  Handgrip strength be measured in both intervention arm and control arm(delayed intervention group.
  Handgrip strength will be measured using Digital Grip Dynamometer TKK5401. Based on the criteria suggested by the Asian Working Group for Sarcopenia, handgrip strength was categorized into two groups: low handgrip strength, < 28 kg for male and < 18 kg for female; and normal handgrip strength, ≥ 28 kg for male and ≥ 18 kg for female
Body composition and handgrip strength | Delayed intervention group : 1) Baseline 2) Pre-evaluation (before exercise program), 3) Post-evaluation ( after 6-week exercise program), 4) long-term evaluation ( after 6months of exercise program)
  Body composition and handgrip strength be measured in both intervention arm and control arm(delayed intervention group).
  Handgrip strength be measured in both intervention arm and control arm(delayed intervention group.
  Handgrip strength will be measured using Digital Grip Dynamometer TKK5401. Based on the criteria suggested by the Asian Working Group for Sarcopenia, handgrip strength was categorized into two groups: low handgrip strength, < 28 kg for male and < 18 kg for female; and normal handgrip strength, ≥ 28 kg for male and ≥ 18 kg for female

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine Division of Pulmonology, Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided